CLINICAL TRIAL: NCT03320499
Title: Impact on Patient Satisfaction About Realization of Ultrasound Dopplers at the Bed
Status: Withdrawn | Type: Observational
Why Stopped: The principal investigator decided to stop the study.
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: SAPHODOPPLER
Record Dates: First submitted 2017-10-16; First posted 2017-10-25 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Ultrasound Doppler

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- echo doppler at the bed
  Interventions: Procedure: echo doppler at the bed
- echo doppler in the vascular exploration platform
  Interventions: Procedure: echo doppler in the vascular exploration platform

INTERVENTIONS:
Procedure: echo doppler at the bed — we practise the echo doppler at the patient 's bed
  Groups: echo doppler at the bed
Procedure: echo doppler in the vascular exploration platform — as usual , practising echo doppler in the medical platform
  Groups: echo doppler in the vascular exploration platform

SUMMARY:
Organisation and logistic about realisation of vascular doppler ultrasound is something very eclectic . Need to shift patient from their bed , long waiting time and the effect on the hospital cost.

That's why vascular yard aim to practise these doppler ultrasound directly in the patients' room in the bed.

And like that evaluate the patient's satisfaction of this kind of coverage.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized in vascular yard
* indication of ultrasound doppler
* accept to participate

Exclusion Criteria:

* refuse to participate
* without ultrasound doppler indication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients hospitalized in vascular yard of GHPSJ
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
score of a satisfaction questionnaire | 24 hours
  in the current practice every patient fill up a questionnaire named SAPHORA to evaluate their satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: PRIOLLET Pascal, MD, Study Director — GHPSJ